CLINICAL TRIAL: NCT02940288
Title: Acupuncture for Postoperative Analgesia in Laparoscopic Surgery
Acronym: Acu-Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Yanire Nieves, Instructor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB00086184
Record Dates: First submitted 2016-10-19; First posted 2016-10-20 (Estimated); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Surgery
MeSH Terms: interventions — Acupuncture, Ear

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Participants will be randomized to receive bilateral auricular acupuncture for postoperative pain.
  Interventions: Other: Auricular Acupuncture
- Control (Sham Comparator): Participants will be randomized to receive bilateral sham acupuncture.
  Interventions: Other: Sham Acupuncture

INTERVENTIONS:
Other: Auricular Acupuncture — Participants will receive bilateral auricular acupuncture using the Battlefield Acupuncture (BFA) protocol while in the Post Analgesia Care Unit (PACU) following laparoscopic surgery. Acupuncture needles will be left in place for 30 minutes.
  Arms: Intervention
Other: Sham Acupuncture — Participants will receive sham acupuncture while in the Post Analgesia Care Unit (PACU) following laparoscopic surgery. During the sham procedure, needles will be inserted bilaterally in five nonspecific ear acupoints. Acupuncture needles will be left in place for 30 minutes.
  Arms: Control

SUMMARY:
Auricular (ear) acupuncture treatment involves placing filiform needles in the ears at particular locations called acupoints. Although the mechanism for acupuncture analgesia is still unclear, it is believed ear acupoints work like reflex points that once stimulated with penetration by a needle have the ability to relieve pain in a different part of the body.

The purpose of this study is to explore the safety and effects of auricular acupuncture therapy on postoperative analgesic consumption and pain scores immediately following laparoscopic surgery.

DETAILED DESCRIPTION:
Auricular acupuncture is a diagnostic and treatment system associated with a somatotopic representation of the homunculus in the ear. This acupuncture technique is similar, in theory, to reflexology where stimulation of a reflex point in the ear is presumed to relieve symptoms in another part of the body. It is hypothesized that this technique works to decrease pain through the reticular formation, the sympathetic and the parasympathetic nervous systems.

The increasing use of laparoscopic surgery has significantly diminished the dosing and duration of postoperative opioid consumption compared with open surgery. However, adverse events related with opioid use (nausea & vomiting, pruritus, urinary retention, sedation) may cause delays in hospital discharge and can be especially problematic for certain sub-sets of high risk patients such as those with obstructive sleep apnea or prior histories of addiction. Investigators hypothesize that auricular acupuncture using the Battlefield Acupuncture Protocol will decrease opioid consumption and postoperative pain after laparoscopic surgery with minimal or no adverse events.

The primary aim of this study is to assess the effects of the BFA protocol on postoperative analgesic consumption and the secondary aims are to assess pain scores and time to discharge from Post Anesthesia Care Unit following laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic surgery for cholecystectomy, hysterectomy or hernia repair
* Patients naïve to acupuncture

Exclusion Criteria:

* Pregnancy
* Bleeding disorder
* Anticoagulant medications
* Involuntary movement disorders/Seizure disorders
* Local auricular infection, loss of skin integrity or significant deformation
* History of opioid medication use or dependence
* Hemodynamic or immunocompromised status
* History of syncope with venipuncture
* Unable to understand the consent form or how to use the VAS-100
* Prosthetic cardiac valves
* Patients will be withdrawn from the study if surgery time exceeds 90 minutes or the laparoscopic procedure turned into an open surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09; Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
Time to First Analgesic Request | Post Surgery (Up to 30 minutes)
  The time to request for analgesia will be collected from the participant's postoperative anesthesia care unit (PACU) records.
Total Amount of Postoperative Pain Medication | Post Surgery (Up to 2 Hours)
  The total amount of pain medication taken up to two hours post surgery will be collected from the participant's postoperative anesthesia care unit (PACU) records.
Pain Intensity assessed by the Visual Analog Scale (VIS) | Post Surgery (Up to 2 Hours)
  Pain intensity will be recorded using the modified 100mm visual analog scale. This scale rates pain from 0 to 100 with 0 meaning no pain at all and 100 is the most severe pain.

SECONDARY OUTCOMES:
Time to Discharge | Post Surgery (Up to 2 Hours)
  Time to discharge from the postoperative anesthesia care unit (PACU) will be collected from the participant's record.

CONTACTS AND LOCATIONS:
Overall Officials: Yanire Nieves, MD, Principal Investigator — Emory University
Locations (1):
- Atlanta Veterans Affairs (VA) Medical Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garimella V, Cellini C. Postoperative pain control. Clin Colon Rectal Surg. 2013 Sep;26(3):191-6. doi: 10.1055/s-0033-1351138. PMID 24436674
- [Background] Sun Y, Gan TJ, Dubose JW, Habib AS. Acupuncture and related techniques for postoperative pain: a systematic review of randomized controlled trials. Br J Anaesth. 2008 Aug;101(2):151-60. doi: 10.1093/bja/aen146. Epub 2008 Jun 2. PMID 18522936
- [Background] Gori L, Firenzuoli F. Ear acupuncture in European traditional medicine. Evid Based Complement Alternat Med. 2007 Sep;4(Suppl 1):13-6. doi: 10.1093/ecam/nem106. PMID 18227925
- [Background] Han JS. Acupuncture and endorphins. Neurosci Lett. 2004 May 6;361(1-3):258-61. doi: 10.1016/j.neulet.2003.12.019. PMID 15135942
- [Background] Usichenko TI, Dinse M, Hermsen M, Witstruck T, Pavlovic D, Lehmann C. Auricular acupuncture for pain relief after total hip arthroplasty - a randomized controlled study. Pain. 2005 Apr;114(3):320-327. doi: 10.1016/j.pain.2004.08.021. PMID 15777857
- [Background] Crespin DJ, Griffin KH, Johnson JR, Miller C, Finch MD, Rivard RL, Anseth S, Dusek JA. Acupuncture provides short-term pain relief for patients in a total joint replacement program. Pain Med. 2015 Jun;16(6):1195-203. doi: 10.1111/pme.12685. Epub 2015 Jan 13. PMID 25586769
- [Background] Goertz CM, Niemtzow R, Burns SM, Fritts MJ, Crawford CC, Jonas WB. Auricular acupuncture in the treatment of acute pain syndromes: A pilot study. Mil Med. 2006 Oct;171(10):1010-4. doi: 10.7205/milmed.171.10.1010. PMID 17076456
- [Background] Han JS, Tang J, Ren MF, Zhou ZF, Fan SG, Qiu XC. Central neurotransmitters and acupuncture analgesia. Am J Chin Med. 1980 Winter;8(4):331-48. doi: 10.1142/s0192415x80000311. PMID 6113756
- [Background] Grube T, Uhlemann C, Weiss T, Meissner W. [Influence of acupuncture on postoperative pain, nausea and vomiting after visceral surgery : a prospective, randomized comparative study of metamizole and standard treatment]. Schmerz. 2009 Aug;23(4):370-6. doi: 10.1007/s00482-009-0798-1. German. PMID 19513760
- [Background] Usichenko TI, Kuchling S, Witstruck T, Pavlovic D, Zach M, Hofer A, Merk H, Lehmann C, Wendt M. Auricular acupuncture for pain relief after ambulatory knee surgery: a randomized trial. CMAJ. 2007 Jan 16;176(2):179-83. doi: 10.1503/cmaj.060875. PMID 17224599
- [Background] Usichenko TI, Hermsen M, Witstruck T, Hofer A, Pavlovic D, Lehmann C, Feyerherd F. Auricular Acupuncture for Pain Relief after Ambulatory Knee Arthroscopy-A Pilot Study. Evid Based Complement Alternat Med. 2005 Jun;2(2):185-189. doi: 10.1093/ecam/neh097. Epub 2005 May 11. PMID 15937559
- [Background] Tan JY, Molassiotis A, Wang T, Suen LK. Adverse events of auricular therapy: a systematic review. Evid Based Complement Alternat Med. 2014;2014:506758. doi: 10.1155/2014/506758. Epub 2014 Nov 10. PMID 25435890
- [Background] Lewith GT, Machin D. On the evaluation of the clinical effects of acupuncture. Pain. 1983 Jun;16(2):111-127. doi: 10.1016/0304-3959(83)90202-6. PMID 6348651
- [Background] Zhang CS, Yang AW, Zhang AL, May BH, Xue CC. Sham control methods used in ear-acupuncture/ear-acupressure randomized controlled trials: a systematic review. J Altern Complement Med. 2014 Mar;20(3):147-61. doi: 10.1089/acm.2013.0238. Epub 2013 Oct 19. PMID 24138333
- [Background] Bohnert AS, Ilgen MA, Galea S, McCarthy JF, Blow FC. Accidental poisoning mortality among patients in the Department of Veterans Affairs Health System. Med Care. 2011 Apr;49(4):393-6. doi: 10.1097/MLR.0b013e318202aa27. PMID 21407033
- [Background] Compton WM, Jones CM, Baldwin GT. Relationship between Nonmedical Prescription-Opioid Use and Heroin Use. N Engl J Med. 2016 Jan 14;374(2):154-63. doi: 10.1056/NEJMra1508490. No abstract available. PMID 26760086
- See also: Prescription Opioids and Heroin — https://www.drugabuse.gov/publications/research-reports/relationship-between-prescription-drug-abuse-heroin-use/introduction
- See also: Design and Rationale of a Comparative Effectiveness Study to Evaluate Two Acupuncture Methods for the Treatment of Headaches Associated with Traumatic Brain Injury — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3579199/